CLINICAL TRIAL: NCT03162601
Title: C-arm Computed Tomography Scan Image Quality in Patients With Neurovascular Diseases: Observational Study
Brief Title: C-arm Computed Tomography Scan Image Quality in Patients With Neurovascular Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Vitor Pereira, Associate Professor of Radiology and Surgery, University Health Network, Toronto
Other Study IDs: TWH-Version 2.0 Sept 28 2016
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Endovascular Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurovascular: Patients to receive percutaneous neurovascular intervention
  Interventions: Procedure: Neurovascular percutaneous intervention

INTERVENTIONS:
Procedure: Neurovascular percutaneous intervention — Patient will receive one extra CACT scan while they are receiving percutaneous neurovascular intervention.

SUMMARY:
With new developments that have taken place in the optimization of C-arm computed tomography (CACT) image acquisition and reconstruction, CACT image quality will be better than current standard-of-care CACT scan techniques used for neurovascular patients referred to endovascular treatment or diagnosis. As such, novel acquisition, filtration, artifact reduction and reconstruction techniques will be evaluated against the standard-of-care CACT approach.

DETAILED DESCRIPTION:
This prospective observational study aims to enroll 50 patients diagnosed with various neurovascular conditions with the goal to compare the image quality of new types of head C-arm computed tomography (CACT) image scans with standard CACT scans, and also to compare these novel scans with standard CT scan image quality. These new scans use novel acquisition, filtration and reconstruction techniques compared to the standard-of-care CACT scans being used in the neuroangiography suite at the present time. Patient selection will be based on a suitability of patients for neuro-endovascular interventions in the neuroangiography suite. All research related activities will be done by study team members. The study patients are expected to follow their routine treatment schedule with the exception of 1 extra CACT scan while patient is receiving their standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is suitable for an endovascular treatment in the neuro-angiography suite.
2. Subject or subject's legally authorized representative has signed an institutionally approved research informed consent form.
3. Subject ≥ 18 years old.

Exclusion Criteria:

1. Subject or subject's legally authorized representative is unable or unwilling to consent to the study.
2. Subject had prior significant or severe allergy to intra-arterial contrast medium uncontrolled by pre-procedure medications.
3. Subject with documented contrast injection contraindication due to severe kidney disease or allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with neurovascular diseases and conditions that are amenable to endovascular treatment in the neuro-angiography suite.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with improved new CACT image quality compared to standard CACT based on a 5-point Likert scale | 1 year
  To achieve a brain parenchyma image quality with CACT using novel acquisition, filtration, artifact reduction and reconstruction techniques that is better than current standard-of-care CACT approaches, based on a 5-point Likert scoring scale questionnaire for each patient.

SECONDARY OUTCOMES:
Number of participants with a CACT image quality at the same level or better as standard CT based on a 5-point Likert scale | 1 year
  Achieve CACT image quality equivalent to or better than standard CT scans (if available) in patients with neurovascular diseases or conditions. This comparison will be done based on a 5-point Likert scoring scale questionnaire for each patient.
Number of participants with improved or equivalent contrast-to-noise ratio using new CACT vs. standard CT scans | 1 year
  Contrast-to-noise ratio (unitless quantity) equivalent or higher in new CACT images compared to standard CT images, measured using regions of interest in image processing software.
Number of participants with improved contrast-to-noise ratio using new CACT vs. standard CACT | 1 year
  Contrast-to-noise ratio (unitless quantity) higher in new CACT images compared to standard CACT images, measured using regions of interest in image processing software.

CONTACTS AND LOCATIONS:
Overall Officials: Vitor Pereira, MD, Principal Investigator — Associate Professor of Radiology and Surgery
Locations (1):
- Toronto Western Hospital - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No